CLINICAL TRIAL: NCT00519506
Title: A Phase II Study to Evaluate the Efficacy of Anti-Fibrin Humanized Monoclonal Antibody(DI-DD3B6/22-80B3) Fab' Fragment (ThromboView®) Conjugated With Technetium-99m in the Detection of Pulmonary Emboli
Brief Title: A Phase II Study to Evaluate the Efficacy of ThromboView® in the Detection of Pulmonary Emboli
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agen Biomedical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAN/US-002-II-PE
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Acute Pulmonary Embolism
Keywords: Pulmonary Embolism; PE
MeSH Terms: conditions — Pulmonary Embolism | interventions — thromboview

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ThromboView — Radiopharmaceutical, single dose, of the diagnosis of venous thromboembolism

SUMMARY:
The aim of the study is to determine the diagnostic accuracy of 99mTc ThromboView® SPECT imaging for the detection of acute pulmonary embolism (PE) in patients for whom there is a moderate to high clinical suspicion for PE.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent by the subject to participate in the study.
2. Moderate to high pre-test probability of acute pulmonary embolism.
3. Positive D-dimer.
4. Onset of PE symptoms occurring within the last seven days.
5. Aged 18 years or older.
6. Women of childbearing potential must have a negative serum pregnancy test (β-hCG) result at the time of enrollment into the study. Both male and female participants must agree to use effective contraception for the first 30 days after administration of 99mTc ThromboView®.

Exclusion Criteria:

1. The subject is unwilling or unable to provide written informed consent.
2. Allergy or other contraindication to intravenous iodinated contrast media.
3. Prior exposure to murine, chimeric or humanized antibodies.
4. Illicit intravenous drug use in the past 12 months.
5. Administration of therapeutic radioiodine in the past 6 months.
6. Life expectancy less than 90 days.
7. Previous participation in the current study.
8. Current enrollment in a clinical trial involving any other investigational agent.
9. Subject is unsuitable for SPECT scanning at the study Investigator's discretion (e.g. residual detectable radioactivity within the lungs due to prior imaging studies or treatment, preceding planned administration of 99mTc ThromboView®).
10. Inability to perform CTPA or 99mTc ThromboView imaging, for any reason.
11. Renal dysfunction: calculated creatinine clearance < 30 mL/min.
12. Hepatic dysfunction: serum transaminases ≥ 3 x upper limit of normal range.
13. Hepatic dysfunction: subject has history of chronic or currently active liver disease.
14. Current pregnancy or lactation or conception intended within three months of enrollment.
15. Subject is unsuitable for the study at the study Investigator's discretion. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Provide estimates of the sensitivity of 99mTc ThromboView® in subjects with confirmed PE, as determined by computed tomographic pulmonary angiography (CTPA) and the specificity of 99mTc ThromboView® in subjects with PE excluded by CTPA | June 2008

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morris, MD, Principal Investigator — UCSD Medical Center
Locations (6):
- United States (4):
  - UC Davis Medical Center, Sacramento, California
  - UCSD Medical Center, San Diego, California
  - Henry Forde Hospital, Detroit, Michigan
  - Washington University School of Medicine at St. Louis, St Louis, Missouri
- Canada (2):
  - McMaster University Medical Center, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario

REFERENCES:
- [Derived] Morris TA, Gerometta M, Yusen RD, White RH, Douketis JD, Kaatz S, Smart RC, Macfarlane D, Ginsberg JS. Detection of pulmonary emboli with 99mTc-labeled anti-D-dimer (DI-80B3)Fab' fragments (ThromboView). Am J Respir Crit Care Med. 2011 Sep 15;184(6):708-14. doi: 10.1164/rccm.201104-0624OC. Epub 2011 Jun 16. PMID 21680946